CLINICAL TRIAL: NCT02239445
Title: Intranasal Dexmedetomidine VS Oral Chloral Hydrate for Rescue Sedation During Magnetic Resonance Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Wenhua Zhang, Bureau of Health of Guangzhou, Guangzhou Women and Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: WZhang
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Administration Related Reaction; Failed Moderate Sedation During Procedure; Chloral Hydrate Adverse Reaction

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- chloral hydrate group (Active Comparator): chloral hydrate 0.25 mg/kg oral solution diluted with oral syrup to 5 ml and 0.2 mL intranasal placebo (normal saline)
  Interventions: Drug: chloral hydrate Group
- low dose dexmedetomidine Group (Experimental): Group L received intranasal dexmedetomidine at 1mcg/kg and 5 ml oral syrup
  Undiluted preservative-free dexmedetomidine (AiBeiNing; Jiang Su Heng Rui Medicine Co. Ltd, Jiangsu Province, China) was prepared in a concentration of 100mcg/ml and dripped into both nostrils using a 1 mL syringe with the child in the Supine position.
  Interventions: Drug: low dose dexmedetomidine group
- high dose dexmedetomidine group (Experimental): Group H received intranasal dexmedetomidine at 2mcg/kg and 5 ml oral syrup
  Undiluted preservative-free dexmedetomidine (AiBeiNing; Jiang Su Heng Rui Medicine Co. Ltd, Jiangsu Province, China) was prepared in a concentration of 100mcg/ml and dripped into both nostrils using a 1 mL syringe with the child in the Supine position.
  Interventions: Drug: high dose dexmedetomidine group

INTERVENTIONS:
Drug: chloral hydrate Group — chloral hydrate 0.25 mg/kg oral solution diluted with oral syrup to 5 ml and 0.2 mL intranasal placebo (normal saline)
  Arms: chloral hydrate group
Drug: low dose dexmedetomidine group — Group L received intranasal dexmedetomidine at 1mcg/kg and 5 ml oral syrup
  Other Names: AiBeiNing
  Arms: low dose dexmedetomidine Group
Drug: high dose dexmedetomidine group — Group H received intranasal dexmedetomidine at 2mcg/kg and 5 ml oral syrup
  Other Names: AiBeiNing
  Arms: high dose dexmedetomidine group

SUMMARY:
The purpose of this investigation was to test the hypothesis that intranasal dexmedetomidine is as effective as second dose of oral chloral hydrate for rescue sedation in infant age between 1 and 6 months who were not adequately sedated following initial dose of chloral hydrate.

ELIGIBILITY:
Inclusion Criteria:

* 160 children of ASA physical status I or II, aged between 1 and 6 months, failed chloral hydrate sedation during MRI scanning

Exclusion Criteria:

* known allergy or hypersensitive reaction to dexmedetomidine or CH, organ dysfunction, pneumonia, acute upper respiratory airway inflammation, preterm, cardiac arrhythmia or and congenital heart disease.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
successful rescue sedation rate | up to 1 hours after MRI scaning
  Sedation status was evaluated by a attending anesthesiologists every 5-10 min with a 6-point sedation scale, which was modified from the Observer Assessment of Alertness and Sedation Scale (MOAA/S; Table 1).
  successful sedation was defined as an MOAA/S of between 0 and 3

SECONDARY OUTCOMES:
sedation induction time | up to 30 min after rescue drug administration
  Successful sedation was defined as an MOAA/S of between 0 and 2, and sedation induction time was defined as the time from rescue drug administration to the onset of satisfactory sedation
  0 Does not respond to a noxious stimulus
  1. Does not respond to mild prodding or shaking
  2. Responds only after mild prodding or shaking
  3. Responds only after name is called loudly orrepeatedly
  4. Lethargic response to name spoken in normal tone
  5. Appears asleep, but responds readily to namespoken in normal tone
  6. Appears alert and awake, responds readily to namespoken in normal tone
Wake -up time | up to 4 hours after rescue drug administration
  Children were classified as awake if the MOAA/S was between 4 and 6. Wake -up time was defined as the time from successful sedation until the time that the child awoke

OTHER OUTCOMES:
non-invasive systolic blood pressure | baseline, before and 15 , 30, 60, 75, 90 min after rescue drug administration
  changes in the non-invasive systolic blood pressure at the baseline, before and 15 , 30, 60, 75, 90 min after rescue drug administration
heart rate | baseline, before and 15 , 30, 60, 75, 90 min after rescue drug administration
  changes in heart rates at the baseline, before and 15 , 30, 60, 75, 90 min after rescue drug administration
Oxyhemoglobin desaturation | baseline and four hours after rescue medicine administration
  Significant Oxyhemoglobin desaturation was defined as<94%

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Anesthesiology of Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong

REFERENCES:
- [Derived] Fong CY, Lim WK, Li L, Lai NM. Chloral hydrate as a sedating agent for neurodiagnostic procedures in children. Cochrane Database Syst Rev. 2021 Aug 16;8(8):CD011786. doi: 10.1002/14651858.CD011786.pub3. PMID 34397100
- [Derived] Zhang W, Wang Z, Song X, Fan Y, Tian H, Li B. Comparison of rescue techniques for failed chloral hydrate sedation for magnetic resonance imaging scans--additional chloral hydrate vs intranasal dexmedetomidine. Paediatr Anaesth. 2016 Mar;26(3):273-9. doi: 10.1111/pan.12824. Epub 2015 Dec 30. PMID 26714442
- [Derived] Miller J, Xue B, Hossain M, Zhang MZ, Loepke A, Kurth D. Comparison of dexmedetomidine and chloral hydrate sedation for transthoracic echocardiography in infants and toddlers: a randomized clinical trial. Paediatr Anaesth. 2016 Mar;26(3):266-72. doi: 10.1111/pan.12819. Epub 2015 Nov 30. PMID 26616644